CLINICAL TRIAL: NCT06812247
Title: Therapy Dog Visits for Patients Hospitalized With Traumatic Injuries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Boston Medical Center Healing Pups Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H45457
Record Dates: First submitted 2025-02-01; First posted 2025-02-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Trauma Injury; Depression; Anxiety; Anger; Pain
Keywords: Therapy dogs; Healing pups; Animal assisted therapy (AAT); Traumatic injuries recovery
MeSH Terms: conditions — Accidental Injuries; Depression; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy dog visits (Experimental): Participants randomized into this arm will receive visits from a therapy dog and their handler during hospitalization.
  Interventions: Other: Therapy dog visits
- Dog handler visits (Active Comparator): Participants randomized into this arm will receive visits from a dog handler during hospitalization.
  Interventions: Other: Dog handler visits

INTERVENTIONS:
Other: Therapy dog visits — 2-3 ten-minute visits by a trained therapy dog and the dog's handler
  Arms: Therapy dog visits
Other: Dog handler visits — 2-3 ten-minute visits by a dog handler
  Arms: Dog handler visits

SUMMARY:
Animal assisted therapy (AAT) with dogs has been shown to be beneficial for a wide range of patients with both acute and chronic illnesses, including spinal cord injuries, heart failure, myocardial infarctions, strokes, cancer, post-traumatic stress disorder, and depression. Studies have also demonstrated that even in healthy adults, the presence of dogs is associated with physiologic changes such as increased pain threshold, decreased blood pressure, and decreased heart rate. However, few studies have investigated the role of AAT in the post-operative course in adults. This study will investigate the impact of therapy dog visits on pain and anxiety scores for trauma patients at Boston Medical Center (BMC).

DETAILED DESCRIPTION:
This study will be a randomized control design. Within 48 hours of admission, the study team will approach eligible patients admitted to the inpatient trauma service to discuss the study and obtain informed consent from patients expected to be admitted for 3-7 days. Consenting patients will be randomized to either a) participate in 2-3 ten-minute dog visits or b) receive 2-3 ten-minute visits with a handler alone. Within 24 hours after the last anticipated study visit, a member of the study team will administer a survey to assess participants' pain, depression, anxiety, mood, and emotional quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Trauma and Acute Care Surgery (TACS) service following a trauma
* English or Spanish speaking
* Able to provide informed consent

Exclusion Criteria:

* Fear of dogs, allergy to dogs
* Immunocompromised
* Contact precautions
* Delirious, intubated, or otherwise unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Participants' pain assessed with a numeric analog score | 24 hours after the last study visit
  The visual analog score ranges from 0 to 10 where 0= no pain and 10 worst pain (5= moderate pain).
Participants' pain assessed with pictures of facial expressions | 24 hours after the last study visit
  The 6 facial pictorial expressions range from 0 to 10 where 0 is a face with a broad smile and 10 is a very sad face with tears.
Depression assessed by the Brief Mood Survey | 24 hours after the last study visit
  There are 5 questions related to feeling depressed in the Brief Mood Survey with five potential responses of- 'Not at all', 'Somewhat', 'Moderately', 'A lot', and 'Extremely'. The range of scores for each of the 5 questions is 0 to 4, with a summed total score of 0 to 20 for the domain and higher scores are associated with feeling more depressed.
Anxiety assessed by the Brief Mood Survey | 24 hours after the last study visit
  There are 5 questions related to feeling anxious in the Brief Mood Survey with five potential responses of- 'Not at all', 'Somewhat', 'Moderately', 'A lot', and 'Extremely'. The range of scores for each of the 5 questions is 0 to 4, with a summed total score of 0 to 20 for the domain, and higher scores are associated with feeling more anxious.
Anger assessed by the Brief Mood Survey | 24 hours after the last study visit
  There are 5 questions related to feeling angry in the Brief Mood Survey with five potential responses of- 'Not at all', 'Somewhat', 'Moderately', 'A lot', and 'Extremely'. The range of scores for each of the 5 questions is 0 to 4, with a summed total score of 0 to 20 for the domain, and higher scores are associated with feeling more angry.

SECONDARY OUTCOMES:
Emotional quality of life now | 24 hours after the last study visit
  The Emoqol-100 will be used to assess emotional quality of life. It is one question, 'How is your emotional quality of life now, with 100 being perfect and 0 being the worst imaginable?' Higher numbers are associated with a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Sanchez, MD MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Trauma Inpatient Service, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No